CLINICAL TRIAL: NCT06903065
Title: A Phase Ib, Multicenter, Open-Label, Single-Arm Study to Assess the Safety, Pharmacokinetics, and Activity of RO7790121 in Patients With Advanced MASH Liver Fibrosis
Brief Title: A Study to Assess the Safety, Pharmacokinetics, and Activity of RO7790121 in Participants With Advanced MASH Liver Fibrosis
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CC45687
Record Dates: First submitted 2025-03-18; First posted 2025-03-30 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: MASH

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- RO7790121 (Experimental): Particiapants will receive RO7790121 via intravenous (IV) infusion followed by subcutaneous (SC) injections.
  Interventions: Drug: RO7790121

INTERVENTIONS:
Drug: RO7790121 — Participants will be administered RO7790121 via IV infusion on Day 1, and Weeks 2, 6 and 10. Participants will then be administered RO7790121 SC injections every four weeks (Q4W) from week 14 up to and including Week 50.
  Other Names: PF-06480605; RVT-3101; RG6631

SUMMARY:
The purpose of this study is to assess the safety, pharmacokinetics (PK), pharmacodynamics (PD), immunogenicity and activity of RO7790121 in participants with advanced metabolic dysfunction-associated steatohepatitis (MASH) fibrosis.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index within the range of >= 25 and <=45 kilograms per square meter (kg/m^2)
* MASH with fibrosis score of F3 or F4 confirmed by transient elastography measurement >=12.0 kPa and <=25.0 kPa
* Agreement to adhere to the contraception requirements

Exclusion Criteria:

* Weight gain or loss >5% in the 3 months prior to baseline or >10% in the 6 months prior to baseline
* Bariatric surgery within 1 year prior to baseline
* Current signs or prior history of decompensated liver disease
* Complications or clinical evidence of portal hypertension
* Lack of peripheral venous access
* Other causes of liver disease based on medical history and/or centralized review of liver histology
* History of liver transplantation
* Current or prior history of hepatocellular carcinoma (HCC)
* Uncontrolled hypertension
* Concomitant Type 1 diabetes, or Type 2 diabetes with HbA1c >10%
* History of malignancy within 5 years prior to screening, with the exception of malignancies with a negligible risk of metastasis or death
* Current, significant alcohol consumption or a history of significant alcohol consumption for a period of more than 3 consecutive months any time within 1 year prior to screening
* Initiation of a medication of an antidiabetic, weight loss, lipid-modifying or anti-depressant drug class
* Active tuberculosis requiring treatment within the 12 months prior to baseline
* History of organ transplant

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-04-14 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of Participants with Adverse Events (AEs) | Up to Week 52 after Baseline

SECONDARY OUTCOMES:
Change from Baseline in Liver Stiffness | Baseline to Week 52
  Liver stiffness will be measured by transient elastography (FibroScan® or FibroTouch®) and indicated in kilopascals (kPa).
Change from Baseline in Serum Levels of Propeptide of Type lll Collagen (Pro-C3) | Baseline to Week 52
Change from Baseline in Serum Enhanced Liver Fibrosis (ELF) Test | Baseline to Week 52
Change from Baseline in Fibro-inflammation | Baseline to Weeks 52
  Fibro-inflammation will be measured using magnetic resonance imaging iron-corrected T1 mapping (MRI cT1).
Pre-dose Concentrations of RO7790121 | Weeks 0, 2, 6, 10, 14, 26, and 38
Maximum Concentration (Cmax) of RO7790121 | Weeks 0, 2, 6, 10, 52 and 62
Minimum Concentration (Cmin) of RO7790121 | Weeks 0, 2, 6, 10, 52 and 62

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (24):
- United States (14):
  - Adobe Clinical Research, LLC, Tucson, Arizona
  - Gastro Health Research - Miami, Miami, Florida
  - Gastrointestinal Specialists of Georgia, PC, Marietta, Georgia
  - Delta Research Partners, LLC (Bastrop), Bastrop, Louisiana
  - Jubilee Clinical Research NV, LLC, Las Vegas, Nevada
  - Innovative Clinical Research, Clarksville, Tennessee
  - Gastroenterology Center of the MidSouth PC, Cordova, Tennessee
  - Pinnacle Clinical Research - Austin, Austin, Texas
  - Bellaire Clinical Research, LLC, Bellaire, Texas
  - DHR Health Institute for Research and Development, Edinburg, Texas
  - Pinnacle Clinical Research Georgetown, Georgetown, Texas
  - Pinnacle Clinical Research, PLLC, San Antonio, Texas
  - GI Alliance, Southlake, Texas
  - GI Alliance, Bellevue, Washington
- Mexico (8):
  - CIMAB S.A. de C.V., Torreón, Coahuila
  - Centro de Investigacion Clinica y Medicina Traslacional CIMeT, Guadalajara, Jalisco
  - Hospital General de Occidente SSJ, Zapopan, Jalisco
  - Inovacion y Desarrollo en ciencias de la salud, Ciudad de Mxico, Mexico CITY (federal District)
  - Centro de Investigacion y Gastroenterologia, Mexico City, Mexico CITY (federal District)
  - Clínica de Enfermedades Crónicas y de Procedimientos Especiales, S.C (CECYPE), Morelia, Michoacán
  - Fundacion Santos Y De La Garza Evia IBP, San Pedro Garza García, Nuevo León
  - Mediadvance Clinical SAPI De CV, Chihuahua City
- Puerto Rico (2):
  - FDI Clinicial Research - Mayaguez, Mayagez
  - Fundacion de Investigacion de Diego, San Juan

IPD SHARING:
Plan to Share IPD: No